CLINICAL TRIAL: NCT06153628
Title: The Effect of Virtual Reality Glasses Applied to Mothers Whose Babies Are in the Neonatal Intensive Care Unit on the Level of Anxiety and the Amount of Breast Milk
Brief Title: The Effect of Virtual Reality Glasses on Anxiety Level and Breast Milk Amount
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mersin University (Other)
Responsible Party: Principal Investigator, Aslı EKER, Dr.Lecturer, Mersin University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Mersin Üniversitesi
Record Dates: First submitted 2023-11-08; First posted 2023-12-01 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-05

CONDITIONS: Anxiety; Amount of Breast Milk
Keywords: Anxiety; Breast milk; Breastfeeding; Premature; Virtual reality glasses
MeSH Terms: conditions — Anxiety Disorders; Breast Feeding; Premature Birth

STUDY DESIGN:
Intervention Model Description: Single-subject quasi-experimental research
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Virtual reality glasses (Experimental): First of all, the "State Anxiety Inventory" will be applied to all women (60 women).Then, milk will be expressed from both breasts once a day (10:00) for the first 3 days and the amount of milk expressed will be recorded in the "Breast Milk Amount Tracking Form". After the first 3 days, all women will be relaxed by watching virtual reality glasses (10 minutes) once a day (10:00 in the morning) for 3 days, and the "State Anxiety Inventory" will be applied at the end of the video. Then, milk will be expressed from both breasts and recorded in the "Breast Milk Amount Tracking Form".
  Interventions: Other: Virtual reality glasses

INTERVENTIONS:
Other: Virtual reality glasses — Videos consisting of nature and undersea images will be played through virtual reality glasses, which the woman wants to watch and can change whenever she wants.

SUMMARY:
Pain, anxiety, nausea, vomiting, etc. In coping with symptoms, virtual reality glasses are recommended as a distraction application. The study was planned to examine the effect of virtual reality glasses applied to mothers whose babies were in the neonatal intensive care unit, on the level of anxiety and the amount of breast milk.

DETAILED DESCRIPTION:
Although milk is expressed early and frequently, milk volume and milk production may be lower in some mothers in the first few weeks.For this reason, pharmacological and non-pharmacological methods have been focused on to increase prolactin secretion and breast milk production in mothers with premature babies. It is emphasized that practices such as breast massage, hot application, nutrition and fluid consumption of the mother, thinking about her baby or looking at her picture, and psychological relaxation during milk expression with a pump increase the amount of milk. It is thought that the mother's stress and anxiety negatively affect the amount of breast milk in preterm births, and that methods that provide relaxation and relief will contribute to breast milk production by reducing stress and anxiety. Pain, anxiety, nausea, vomiting, etc. In coping with symptoms, virtual reality glasses are recommended as a distraction application.

ELIGIBILITY:
Inclusion Criteria:

* Are between the ages of 18-45,
* Those who gave birth at a gestational age of 30 weeks or more,
* whose baby is still in intensive care,
* whose baby has started breastfeeding,
* Giving breast milk to her baby by expressing,
* Not using any medication that will affect milk supply,
* Not diagnosed with a psychiatric disease that will affect breastfeeding in the postpartum period,
* Those who have not had any breast-related surgery before,
* Understands Turkish and can communicate,
* Mothers who sign the Informed Volunteer Consent Form will be included in the research.

Exclusion Criteria:

* Those who are younger than 18 years of age or older than 45 years of age,
* The gestational age is less than 30 weeks,
* whose baby was discharged from intensive care,
* whose baby has not started breastfeeding,
* Those who do not express breast milk to their babies,
* Using medication that will affect milk supply,
* Diagnosed with a psychiatric disease that will affect breastfeeding in the postpartum period,
* Have had any breast-related surgery before,
* Cannot communicate in Turkish,
* Mothers who do not sign the Informed Volunteer Consent Form will not be included in the research.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Since the study was about breastfeeding, only women were included.
Enrollment: 60 (Actual)
Dates: Start 2023-11-02 (Actual); Primary Completion 2024-04-10 (Actual); Study Completion 2024-06-15 (Actual)

PRIMARY OUTCOMES:
State-Anxiety Inventory | Up to 3 Months
  In the Likert-type scale consisting of 20 items, the items are numbered from 1 to 4 (1 means "not at all" and 4 means "completely").The scores obtained from the scale vary between 20 and 80 and there are direct (straight) and reversed expressions in the scale.

SECONDARY OUTCOMES:
Breast Milk Quantity Monitoring Form | Up to 3 Months
  It is a form consisting of 3 parts developed by the researcher to record information about milking date, milking time and milk amount.

CONTACTS AND LOCATIONS:
Locations (1):
- Mersin University, Mersin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kent JC, Geddes DT, Hepworth AR, Hartmann PE. Effect of warm breastshields on breast milk pumping. J Hum Lact. 2011 Nov;27(4):331-8. doi: 10.1177/0890334411418628. PMID 22048756
- [Background] Hill PD, Aldag JC, Chatterton RT. Effects of pumping style on milk production in mothers of non-nursing preterm infants. J Hum Lact. 1999 Sep;15(3):209-16. doi: 10.1177/089033449901500310. PMID 10578798
- See also: World Health Organization Report of the Expert Consultation on the Optimal Duration of Exclusive Breastfeeding. Geneva, World Health Organization 2001, — https://iris.who.int/bitstream/handle/10665/67219/WHO_NHD_01.09.pdf
- See also: Gartner LM, Morton J, Lawrence RA, Naylor AJ, O'Hare D, Schanler RJ et al. American Academy of Pediatrics Section on Breastfeeding. Breastfeeding and the use of human milk. Pediatrics 2005; 115: 496-506 — https://pubmed.ncbi.nlm.nih.gov/15687461/
- See also: American Academy of Family Physicians (AAFP) (2007). Breastfeeding (policy statement). In. Appendix 2: Additional Breastfeeding Considerations 2010; 13-14 — https://www.aafp.org/about/policies/all/breastfeeding-position-paper.html
- See also: World Health Organization. The Global Action Report on Preterm Birth, 2012; 1-126 — https://iris.who.int/bitstream/handle/10665/44864/9789241503433_eng.pdf